CLINICAL TRIAL: NCT07113717
Title: Early Post-operative Discharge of Colorectal Surgical Patients to a Virtual Hospital at Home Model (Post Operative Hospital at Home) - a Clinical Feasibility Study
Brief Title: Post Operative Hospital at Home After Colorectal Surgery
Acronym: POPHaH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nordsjaellands Hospital (Other)
Responsible Party: Principal Investigator, Kristin Julia Steinthorsdottir, Surgeon, ph.d., Nordsjaellands Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 100100100
Record Dates: First submitted 2025-07-07; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Colo-rectal Cancer; Colo-rectal Surgery; Colocolic and Ileocolic Anastomosis; Colon and/or Rectal Resection With Anastomosis for Cancer; Diverticular Disease of Colon; Colon Benign Tumor; Crohn Disease and Ulcerative Colitis; Ileostomy Closure; Stoma Reversal Procedure
Keywords: hospital at home for colorectal surgery; postoperative hospital at home
MeSH Terms: conditions — Colonic Neoplasms; Diverticulosis, Colonic; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: Feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- virtual Hospital at Home (Experimental): participants admittet to virtual Hospital at Home
  Interventions: Other: virtual Hospital at Home

INTERVENTIONS:
Other: virtual Hospital at Home — telemedicine set-up, virtual Hospital at Home

SUMMARY:
The goal of this feasibility study is to investigate whether a virtual Hospital at Home is safe and possible for patients undergoing planned minimally invasive colorectal surgery. The study aims to answer the following main questions:

What are the patient- and next-of-kin-related effects, as well as the clinical and organizational effects, of home-based admission? What are the implementation barriers for a full-scale randomized controlled trial? Participants will follow a standardized protocol for their care befor, during and after surgery. However, the care after surgery will be conducted at home using telemedicine.

DETAILED DESCRIPTION:
Original Title

Feasibility of Early Post-Operative Discharge to a Virtual Hospital at Home Model for Colorectal Surgical Patients.

Purpose

Project context

Enhanced recovery after surgery (ERAS) is an evidence-based approach designed to help patients recover more quickly and safely after surgery( 1) . It is widely implemented in many centres that offer minimally invasive colorectal surgery (CRS) (2,3) . This multimodal approach aims to reduce the physical and psychological stress of surgery, resulting in lower complication rates, shorter hospital stays, and reduced healthcare costs. Continuous efforts are made to implement and evaluate individual components of the ERAS protocol, ensuring that valuable aspects for patients and society are maintained and enhanced, while redundant elements are eliminated ( 1,4,5) . Optimizing all modifiable patient-related factors before surgery and adhering to standardized peri-operative care pathways is essential when striving to not only surgically remove a disease but also to ensure that patients are better off after surgery ( 6-8) .

The key question and original premise for ERAS is: "Why is the patient still in hospital" (5) . With the technical advancements and necessity brought on by the COVID-19 pandemic, a platform for virtual Hospital at Home (vHaH) was founded. Initially started as an admission-avoidance strategy for patients with acute medical conditions the concept evolved into an 'early discharge' hospital at home model and has been implemented by some elective surgical specialities (primarily orthopaedic) (9-10) .

CRS centres across the USA and Europe have been implementing Virtual Hospital or Same-Day discharge (SDD) for selected patients for the last couple of years (11-16) . Retrospective reviews and analyses of data, although inherently biased, have so far shown non-inferiority and suggested superiority regarding patient experience and safety ( 17-21) . A newly published pilot study on remote monitoring after CRC in rural areas showed feasibility and high patient acceptance ( 22) . However, there seem to be unreported barriers to generalized implementation. So far, there is only very limited documented surgical experience from sound research approaches available in the literature. This surgical feasibility study builds on methods previously tested in a medical population at the investigators' institution ( 23) . The findings will inform the development and design of a randomized clinical trial to evaluate the final telemedicine-supported vHaH model for surgical patients.

The overall aim of POPHaH is to implement a telemedicine monitoring and communication model that will enable the safe admission of postoperative patients in their homes.

A hospital based Virtual Surgical Centre (VSC) will be located in the Department of Surgery at Copenhagen University Hospital - North Zealand (NOH), from where medical staff will monitor and communicate with patients admitted at home. Vital parameters and patient-reported outcomes will be collected using a smartphone/tablet-based app. All data will be collected and displayed in real-time at the NOH in the VSC, allowing medical staff to monitor the vHaH patients similarly to in-patients. In addition, daily virtual ward rounds conducted by staff in the VSC and, when relevant, by medical doctors (MDs) from specialities relevant to the patients' illness(es) will ensure close communication and relevant clinical assessments.

This vHaH model is expected to become an integrated part of the hospital postoperative observation repertoire in the Capital Region of Denmark and elsewhere. In this feasibility study, hospitalized patients with surgical conditions will be offered the opportunity to continue their hospital course as a home-based admission.

Study Purpose

The objective of this feasibility study is to investigate and analyze the key factors involved in admitting adult patients undergoing CRS, including cancer surgery, in a vHaH model. The study aims to evaluate the likelihood of successfully completing the vHaH model in this patient group.

It will focus on assessing outcomes related to patients, their next of kin, clinical aspects and organizational dynamics. Additionally, it will examine factors crucial for determining the feasibility of conducting a full-scale randomized controlled trial.

Research Question

What are the patient- and next-of-kin-related effects, as well as the clinical and organisational effects, of home-based admission? What are the implementation barriers for a full-scale randomized controlled trial?

Hypothesis

The investigators hypothesize that early postoperative discharge of selected CRS patients to a telemedicine-supported vHaH model, will be a viable alternative to conventional hospitalization without compromising patient and next-of-kin safety or satisfaction.

Rationale

Virtual Hospital-at-Home (vHaH) following CRS offers numerous advantages. For patients, it promotes a faster return to normal life, encourages postoperative mobilization, reduces the risk of hospital-acquired infections, and allows recovery in the comfort of their own homes with family support. On a societal level, vHaH presents an opportunity to optimize healthcare resources, and addresses challenges posed by centralization and an aging population.

Over the past two decades, the Danish public healthcare system has undergone significant centralization, resulting in fewer, larger hospitals with a reduced bed capacity at both regional and national levels. At the same time, the aging population and increasing prevalence of multimorbidity have placed additional demands on the system. Prioritizing hospital beds without compromising the quality of care is crucial.

Enhanced Recovery After Surgery (ERAS) pathways have demonstrated that postoperative recovery can be efficient and safe within hospitals. Combining ERAS principles with vHaH models, supported by research on patient safety and satisfaction, enables same-day or next-day discharge to a vHaH after CRS for selected patients.

Given that ERAS pathways were originally designed for CRS, and with nearly two decades of experience in this field, together with the clinical and scientific experience from the medical colleagues in the Department of Pulmonology and Infectious Diseases at the investigators' institution, this surgical department is uniquely positioned to pilot the model. Successfully implementing a surgical vHaH program in this patient group could serve as a blueprint for expanding the approach to other abdominal surgical subspecialities and surgical specialities, further enhancing healthcare delivery across the board. The investigators are conducting a feasibility study to thoroughly examine potential barriers to implementing surgical vHaH, including logistical challenges and patient acceptance. This approach is designed to ensure the model's sustainability and adaptability for broader application. Following this, the investigators plan to evaluate its effectiveness through a randomized controlled trial (RCT).

ELIGIBILITY:
Inclusion Criteria:

* Planned minimally invasive (laparoscopic or robot-assisted) CRS
* No epidural analgesia
* No new stoma
* Bleeding < 500 ml
* Actual condition assessed to be clinically stable
* Meeting the Chung score discharge criteria for ambulatory surgery
* Self-reliant or receives sufficient formal care to be care-independent of a primary informal caregiver
* Home-based admission will be located within catchment area of the hospital (according to the official address of the individual)
* Signed informed written and oral consent

Exclusion Criteria:

* Patients who cannot comply with self-assessment
* Improficiency in Danish
* Pregnancy
* Conversion to emergency surgery (uncontrolled perforation of bowel, ileus)
* Complications during surgery warranting in-hospital admission (observation in intensive care unit or close observation from other specialities, e.g. cardiology)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Number of recruited participants | one year
  Recruitment success is defined as 50% of eligible patients

SECONDARY OUTCOMES:
Number of drop-out participants | one year
  retention success is defined by less than 10% drop-outs
Number of protocol deviations | one year
  Percentage of:
  Planned daily video supported ward rounds provided adherence (successful adherence is defined by 95%)
  Planned self-measurements transmitted by patient adherence (successful adherence is defined by 80%)

OTHER OUTCOMES:
Patient related endpoints (surgical complications) | Thirty days after surgery
  Clavien-Dindo classification:
  * Grade I: Minor complications that do not require specific treatment (e.g., antiemetics, antipyretics).
  * Grade II: Complications requiring pharmacological treatment (e.g., antibiotics, blood transfusions).
  * Grade III: Complications requiring surgical, endoscopic, or radiological intervention.
  * IIIa: Without general anesthesia.
  * IIIb: With general anesthesia.
  * Grade IV: Life-threatening complications requiring intensive care.
  * IVa: Single organ dysfunction.
  * IVb: Multi-organ dysfunction.
Patient related endpoints (readmittance rate) | Thirty days after surgery
  Number of readmittances post discharge
Patient related endpoints (Mortality) | Thirty days after surgery
  Mortality (associated)
Patient related endpoints (Quality of recovery) | Thirty days after surgery
  Quality of Recovery-15 (QoR-15) is a short, patient-centered questionnaire designed to assess the quality of recovery after surgery. It is a streamlined version of the longer QoR-40 and includes 15 items that cover five key dimensions of recovery:
  1. Physical Comfort
  2. Emotional State
  3. Psychological Support
  4. Physical Independence
  5. Pain Scoring: Each item is rated on a scale from 0 to 10, with higher scores indicating better recovery. The total score ranges from 0 to 150
Patient related endpoints (Hours out of bed) | From discharge from post-operative care unit to discharge from home-based admission (estimated 2-4 days, up to maximum 14 days). Measured in hours and minutes.
  Hours out of bed, measured by a SENS motion® accelerometric sensor, detailed data about number of steps.
Patient related endpoint (Sleep) | From discharge from post-operative care unit to discharge from home-based admission (estimated 2-4 days, up to maximum 14 days). Measured in hours and minutes, per 24 hours.
  Lenght (in hours) of sleep, measured with SENS motion® accelerometric sensor
Next-of-kin-related endpoints | one year
  Caregiver strain (primary informal caregivers will be invited to explorative interviews to establish factors of importance)
Unscheduled contacts (including virtual) | From discharge from post-operative care unit to discharge from home-based admission (estimated 2-4 days, up to maximum 14 days). .
  Number of unscheduled contacts during admission
Contacts to general practitioner | From discharge from post-operative care unit to discharge from home-based admission (estimated 2-4 days, up to maximum 14 days).
  Number of contacts to general practitioner during home-based admission
Hours in-hospital | From discharge from post-operative care unit to discharge from home-based admission (estimated 2-4 days, up to maximum 14 days).
  Number of in-hospital hours
Outpatient visits | From discharge until 30 days after surgery
  Number of outpatient visits

CONTACTS AND LOCATIONS:
Overall Officials: Kristin J Steinthorsdottir, MD, Ph.d., Principal Investigator — Nordsjaellands Hospital, Surgical Department
Locations (1):
- Department of Surgery, Hillerød, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vu MM, Curfman KR, Blair GE, Shah CA, Rashidi L. Beyond enhanced recovery after surgery (ERAS): Evolving minimally invasive colectomy from multi-day admissions to same-day discharge. Am J Surg. 2023 May;225(5):826-831. doi: 10.1016/j.amjsurg.2023.01.024. Epub 2023 Jan 21. PMID 36697356
- [Background] Nikmanesh P, Arabloo J, Gorji HA. Dimensions and components of hospital-at-home care: a systematic review. BMC Health Serv Res. 2024 Nov 25;24(1):1458. doi: 10.1186/s12913-024-11970-5. PMID 39587580
- [Background] Gustafsson UO, Scott MJ, Schwenk W, Demartines N, Roulin D, Francis N, McNaught CE, MacFie J, Liberman AS, Soop M, Hill A, Kennedy RH, Lobo DN, Fearon K, Ljungqvist O; Enhanced Recovery After Surgery Society. Guidelines for perioperative care in elective colonic surgery: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations. Clin Nutr. 2012 Dec;31(6):783-800. doi: 10.1016/j.clnu.2012.08.013. Epub 2012 Sep 28. PMID 23099039